CLINICAL TRIAL: NCT00166998
Title: The Study of Infrared Imaging on Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701271
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-02

CONDITIONS: Breast Neoplasms
Keywords: Breast neoplasms; diagnosis
MeSH Terms: conditions — Breast Neoplasms; Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Breast cancer can cause focal temperature increase on the breast skin due to vasodilatation mediated by NO secretion from cancer cells. Our study is to evaluate this situation and to assess the diagnostic efficacy of infrared imaging (thermography)on breast cancer.

DETAILED DESCRIPTION:
Malignant breast neoplasms can secrete NO to induce focal vasodilatation and increased blood flow and angiogenesis to the tumor, thus increase the focal temperature, which can be evaluated by breast thermography (infrared imaging). We will evaluate the efficacy of infrared imaging for detection and diagnosis of breast cancer, and if infrared imaging can effectively differentiate malignant from benign breast dieases and the sensitivity, specificity, false-negative rate will also be estimated.

ELIGIBILITY:
Inclusion Criteria:

* normal group: women who has normal mammograms or ultrasound in 6 months abnormal group: women who has suspicious findings on mammograms or ultrasound in recent 6 months

Exclusion Criteria:

* women who don't fit the above inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2005-03; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Jane Wang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Parisky YR, Sardi A, Hamm R, Hughes K, Esserman L, Rust S, Callahan K. Efficacy of computerized infrared imaging analysis to evaluate mammographically suspicious lesions. AJR Am J Roentgenol. 2003 Jan;180(1):263-9. doi: 10.2214/ajr.180.1.1800263. PMID 12490517
- [Derived] Wu LA, Kuo WH, Chen CY, Tsai YS, Wang J. The association of infrared imaging findings of the breast with prognosis in breast cancer patients: an observational cohort study. BMC Cancer. 2016 Jul 27;16:541. doi: 10.1186/s12885-016-2602-9. PMID 27464553
- [Derived] Wang J, Chang KJ, Chen CY, Chien KL, Tsai YS, Wu YM, Teng YC, Shih TT. Evaluation of the diagnostic performance of infrared imaging of the breast: a preliminary study. Biomed Eng Online. 2010 Jan 7;9:3. doi: 10.1186/1475-925X-9-3. PMID 20055999